CLINICAL TRIAL: NCT03324893
Title: 18F-Fluorocholine PET/MRI for the Localization of Parathyroid Adenomas
Brief Title: FCH PET/MRI Parathyroid Localization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-5153
Record Dates: First submitted 2017-10-17; First posted 2017-10-30 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: 18F-fluorocholine; Positron-Emission Tomography; Hyperparathyroidism, Primary
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [F18]-FCH PET/MRI (Experimental): Patients with primary hyperparathyroidism planned for parathyroidectomy
  Interventions: Diagnostic Test: [F-18]-FCH PET/MRI

INTERVENTIONS:
Diagnostic Test: [F-18]-FCH PET/MRI — Subjects will undergo the [F-18]-FCH PET/MRI within three months prior to scheduled parathyroidectomy.
  Other Names: FCH PET/MRI; Fluorine-18 fluorocholine PET/MRI

SUMMARY:
A prospective trial comparing the accuracy of [F-18]-FCH PET/MRI to US and 99mTc-MIBI SPECT/CT for pre-operative parathyroid localization in patients with primary hyperparathyroidism

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biochemically proven primary hyperparathyroidism
* Indication for parathyroidectomy as per institutional guidelines

Exclusion Criteria:

* Contraindication for MRI as per current institutional guidelines.
* Contraindication for Gadolinium injection as per current institutional guidelines.
* Renal failure
* Inability to lie supine for at least 45 minutes.
* Any participant who is pregnant or breastfeeding.
* Participants receiving erythropoietin (i.e. for hemochromatosis; might lead to false negative results due to stimulation of bone marrow metabolism)
* Familial HPT syndromes
* Participant currently being treated with any cytotoxic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Accuracy of [F-18]-FCH PET/MRI in localization of diseased parathyroid gland | 1 month postoperatively
  Value of [F-18]-FCH PET/MRI next to Ultrasound of the Neck and 99mTc-MIBI SPECT/CT in determining which of the four parathyroid glands
  Reference standards:
  * Intra-operative location of the hyper functioning gland by inspection and post-operative pathological confirmation.
  * Determination of biochemical cure per usual standard of care: intraoperative PTH and calcium and PTH postoperatively.

CONTACTS AND LOCATIONS:
Locations (1):
- UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided